CLINICAL TRIAL: NCT05221697
Title: Effect of an Electronic Alert Management System Using Caregivers' Observations and Machine Learning Algorithm to Reduce the Use of Emergency Department Visits and Unplanned Hospitalizations Among Older People
Brief Title: Effect of an ML Electronic Alert Management System to Reduce the Use of ED Visits and Hospitalizations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Presage (Industry)
Collaborators: Assistance Publique Hopitaux De Marseille (Other); Assistance Publique - Hôpitaux de Paris (Other); University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRESAGE_2021-01
Record Dates: First submitted 2022-01-07; First posted 2022-02-03 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Emergencies
Keywords: Emergency Department visits,; machine learning; smartphone
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): PRESAGE Care ATIH + Nurse or GP consultation
  Interventions: Device: PRESAGE CARE
- Control group (No Intervention): usual care

INTERVENTIONS:
Device: PRESAGE CARE — Participants in this arm will be followed by HCA and might benefit from Nurse health interventions
  Arms: Intervention

SUMMARY:
Development, validation and impact of an alert management system using social workers' observations and machine learning algorithms to predict 7-to-14-day alerts for the risk of Emergency Department (ED) Visit and unplanned hospitalization.

Multi-center trial implementation of electronic Home Care Aides-reported outcomes measure system among patients, frail adults >= 65 years living at home and receiving assistance from home care aides (HCA).

DETAILED DESCRIPTION:
On a weekly basis, after home visit, HCAs reported on participants' functional status using a smartphone application that recorded 23 functional items about each participant (e.g., ability to stand, move, eat, mood, loneliness). Predictive system using Machine learning techniques (i.e., leveraging random forest predictors) was developed and generated 7 to 14-day predictive alerts for the risk of ED visit to nurses.

This questionnaire focused on functional and clinical autonomy (ie, activities of daily life), possible medical symptoms (eg, fatigue, falls, and pain), changes in behavior (eg, recognition and aggressiveness), and communication with the HA or their surroundings. This questionnaire is composed of very simple and easy-to-understand questions, giving a global view of the person's condition. For each of the 23 questions, a yes/no answer was requested. Data recorded by HAs were sent in real time to a secure server to be analyzed by our machine learning algorithm, which predicted the risk level and displayed it on a web-based secure medical device called PRESAGE CARE, which is CE marked. Particularly, when the algorithm predicted a high-risk level, an alert was displayed in the form of a notification on the screen to the coordinating nurse of the health care network center of the district. This risk notification was accompanied by information about recent changes in the patients' functional status, identified from the HAs' records, to assist the coordinating nurse in interacting with family caregiver and other health professionals.

In the event of an alert, the coordinating nurse called the family caregiver to inquire about recent changes in the patient's health condition and for doubt removal and could then decide to ask for a health intervention according to a health intervention model developed before the start of the study. In brief, this alert-triggered health intervention (ATHI) consisted of calling the patient's nurse (if the patient had regular home visits of a nurse) or the patient's general practitioner and informing them of a worsening of the patient's functional status and a potential risk of an ED visit or unplanned hospitalization in the next few days according to the eHealth system algorithm. This model of ATHI had been presented and approved by the Agences Régionales de Santé of the regions involved in our study

ELIGIBILITY:
Inclusion Criteria:

* age of 75 yo mini
* receiving the help of a social worker
* patient should give their consent
* patient should had seen their primary care professional within the past 12 months

Exclusion Criteria:

* People with severe dependence (French national instrument, which stratifies dependency level from group iso-resources (GIR) : 1 (very severe dependency) and 2 (severe dependency)

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Unplanned Hospitalization rate | through study completion, an average of 1 year
  Comparison between unplanned hospitalization ratio from 2 randomized groups (intervention and control arms).
  P values <.05 will be considered statistically significant.
Event-free survival (EFS) | through study completion, an average of 1 year
  Comparison average Time for first adverse event between intervention and control groups.
  P values <.05 will be considered statistically significant.
Impact on older adults and relatives' quality of life (European Quality of Life 5 Dimensions and 3 Lines scale) | through study completion, an average of 1 year
  Comparison of the average score of EQ5D-3L quality of life scale (European Quality of Life 5 Dimensions and 3 Lines) between intervention and control groups.
  P values <.05 will be considered statistically significant.
Cost-effectiveness | through study completion, an average of 1 year
  Incremental cost-effectiveness ratio (ICER), QALY. Willingness-to-pay thresholds of €30,000 per quality-adjusted life year (QALY) and €90,000 per QALY were used to define a very cost-effective and cost-effective strategy, respectively

SECONDARY OUTCOMES:
Impact on users : time needed to complete questionnaire | through study completion, an average of 1 year
  Time needed to complete questionnaire (minutes) : a time of less than 2 minutes will be considered acceptable
Intervention rate | through study completion, an average of 1 year
  Part of alert which leads to interventions and intervention time (%). Rate of over 70% is considered acceptable.
Intervention time | through study completion, an average of 1 year
  Mean of the duration between day of alert and day of intervention (in days). A delay of less than 4 days is considered acceptable.
Time needed to analysis patient statut | through study completion, an average of 1 year
  Time needed to analysis patient statut (hours and minutes) : a time of less than 15 minutes by patient will be considered acceptable
Impact on quality of care | through study completion, an average of 1 year
  Positive or very positive impact on quality of care : rate of over 80% is considered acceptable.
Impact on Professional' Relationship and coordination | through study completion, an average of 1 year
  Positive or very positive impact on professionnal relationship and coordination :rate of over 80% is considered acceptable.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Grand Versailles, Le Chesnay
  - Marseille-1, Marseille

IPD SHARING:
Plan to Share IPD: No
anonymized Statistical data will be available

REFERENCES:
- [Background] Clerencia-Sierra M, Calderon-Larranaga A, Martinez-Velilla N, Vergara-Mitxeltorena I, Aldaz-Herce P, Poblador-Plou B, Machon-Sobrado M, Egues-Olazabal N, Abellan-van Kan G, Prados-Torres A. Multimorbidity Patterns in Hospitalized Older Patients: Associations among Chronic Diseases and Geriatric Syndromes. PLoS One. 2015 Jul 24;10(7):e0132909. doi: 10.1371/journal.pone.0132909. eCollection 2015. PMID 26208112
- [Background] Kahn JH, Magauran BG Jr, Olshaker JS, Shankar KN. Current Trends in Geriatric Emergency Medicine. Emerg Med Clin North Am. 2016 Aug;34(3):435-52. doi: 10.1016/j.emc.2016.04.014. PMID 27475008
- [Background] Gasperini B, Cherubini A, Pierri F, Barbadoro P, Fedecostante M, Prospero E. Potentially preventable visits to the emergency department in older adults: Results from a national survey in Italy. PLoS One. 2017 Dec 21;12(12):e0189925. doi: 10.1371/journal.pone.0189925. eCollection 2017. PMID 29267333
- [Background] McCusker J, Verdon J. Do geriatric interventions reduce emergency department visits? A systematic review. J Gerontol A Biol Sci Med Sci. 2006 Jan;61(1):53-62. doi: 10.1093/gerona/61.1.53. PMID 16456194
- [Background] Inglis SC, Clark RA, McAlister FA, Ball J, Lewinter C, Cullington D, Stewart S, Cleland JG. Structured telephone support or telemonitoring programmes for patients with chronic heart failure. Cochrane Database Syst Rev. 2010 Aug 4;(8):CD007228. doi: 10.1002/14651858.CD007228.pub2. PMID 20687083
- [Background] Chen CC, Wang C, Huang GH. Functional trajectory 6 months posthospitalization: a cohort study of older hospitalized patients in Taiwan. Nurs Res. 2008 Mar-Apr;57(2):93-100. doi: 10.1097/01.NNR.0000313485.18670.e2. PMID 18347480
- [Background] Iwashyna TJ, Ely EW, Smith DM, Langa KM. Long-term cognitive impairment and functional disability among survivors of severe sepsis. JAMA. 2010 Oct 27;304(16):1787-94. doi: 10.1001/jama.2010.1553. PMID 20978258
- [Background] Camargo CA Jr, Tsai CL, Sullivan AF, Cleary PD, Gordon JA, Guadagnoli E, Kaushal R, Magid DJ, Rao SR, Blumenthal D. Safety climate and medical errors in 62 US emergency departments. Ann Emerg Med. 2012 Nov;60(5):555-563.e20. doi: 10.1016/j.annemergmed.2012.02.018. PMID 23089089
- [Background] Crane SJ, Tung EE, Hanson GJ, Cha S, Chaudhry R, Takahashi PY. Use of an electronic administrative database to identify older community dwelling adults at high-risk for hospitalization or emergency department visits: the elders risk assessment index. BMC Health Serv Res. 2010 Dec 13;10:338. doi: 10.1186/1472-6963-10-338. PMID 21144042
- [Background] Hu Z, Jin B, Shin AY, Zhu C, Zhao Y, Hao S, Zheng L, Fu C, Wen Q, Ji J, Li Z, Wang Y, Zheng X, Dai D, Culver DS, Alfreds ST, Rogow T, Stearns F, Sylvester KG, Widen E, Ling XB. Real-time web-based assessment of total population risk of future emergency department utilization: statewide prospective active case finding study. Interact J Med Res. 2015 Jan 13;4(1):e2. doi: 10.2196/ijmr.4022. PMID 25586600
- [Background] Takahashi PY, Heien HC, Sangaralingham LR, Shah ND, Naessens JM. Enhanced risk prediction model for emergency department use and hospitalizations in patients in a primary care medical home. Am J Manag Care. 2016 Jul;22(7):475-83. PMID 27442203
- [Background] Denis F, Krakowski I. How Should Oncologists Choose an Electronic Patient-Reported Outcome System for Remote Monitoring of Patients With Cancer? J Med Internet Res. 2021 Sep 9;23(9):e30549. doi: 10.2196/30549. PMID 34499046
- [Background] Bouazza YB, Chiairi I, El Kharbouchi O, De Backer L, Vanhoutte G, Janssens A, Van Meerbeeck JP. Patient-reported outcome measures (PROMs) in the management of lung cancer: A systematic review. Lung Cancer. 2017 Nov;113:140-151. doi: 10.1016/j.lungcan.2017.09.011. Epub 2017 Sep 23. PMID 29110842
- [Background] Schick-Makaroff K, Karimi-Dehkordi M, Cuthbertson L, Dixon D, Cohen SR, Hilliard N, Sawatzky R. Using Patient- and Family-Reported Outcome and Experience Measures Across Transitions of Care for Frail Older Adults Living at Home: A Meta-Narrative Synthesis. Gerontologist. 2021 Apr 3;61(3):e23-e38. doi: 10.1093/geront/gnz162. PMID 31942997
- [Background] Veyron JH, Friocourt P, Jeanjean O, Luquel L, Bonifas N, Denis F, Belmin J. Home care aides' observations and machine learning algorithms for the prediction of visits to emergency departments by older community-dwelling individuals receiving home care assistance: A proof of concept study. PLoS One. 2019 Aug 13;14(8):e0220002. doi: 10.1371/journal.pone.0220002. eCollection 2019. PMID 31408458
- [Background] Huntley AL, Chalder M, Shaw ARG, Hollingworth W, Metcalfe C, Benger JR, Purdy S. A systematic review to identify and assess the effectiveness of alternatives for people over the age of 65 who are at risk of potentially avoidable hospital admission. BMJ Open. 2017 Aug 1;7(7):e016236. doi: 10.1136/bmjopen-2017-016236. PMID 28765132
- [Background] Seibert K, Domhoff D, Bruch D, Schulte-Althoff M, Furstenau D, Biessmann F, Wolf-Ostermann K. Application Scenarios for Artificial Intelligence in Nursing Care: Rapid Review. J Med Internet Res. 2021 Nov 29;23(11):e26522. doi: 10.2196/26522. PMID 34847057
- [Background] Gray JT, Walker A. Avoiding admissions from the ambulance service: a review of elderly patients with falls and patients with breathing difficulties seen by emergency care practitioners in South Yorkshire. Emerg Med J. 2008 Mar;25(3):168-71. doi: 10.1136/emj.2007.050732. PMID 18299372
- [Background] Mason S, O'Keeffe C, Knowles E, Bradburn M, Campbell M, Coleman P, Stride C, O'Hara R, Rick J, Patterson M. A pragmatic quasi-experimental multi-site community intervention trial evaluating the impact of Emergency Care Practitioners in different UK health settings on patient pathways (NEECaP Trial). Emerg Med J. 2012 Jan;29(1):47-53. doi: 10.1136/emj.2010.103572. PMID 22186262
- [Background] Mason S, Knowles E, Colwell B, Dixon S, Wardrope J, Gorringe R, Snooks H, Perrin J, Nicholl J. Effectiveness of paramedic practitioners in attending 999 calls from elderly people in the community: cluster randomised controlled trial. BMJ. 2007 Nov 3;335(7626):919. doi: 10.1136/bmj.39343.649097.55. Epub 2007 Oct 4. PMID 17916813
- [Background] Soril LJ, Leggett LE, Lorenzetti DL, Noseworthy TW, Clement FM. Reducing frequent visits to the emergency department: a systematic review of interventions. PLoS One. 2015 Apr 13;10(4):e0123660. doi: 10.1371/journal.pone.0123660. eCollection 2015. PMID 25874866
- [Background] Belmin J, Auffray JC, Berbezier C, Boirin P, Mercier S, de Reviers B, Golmard JL. Level of dependency: a simple marker associated with mortality during the 2003 heatwave among French dependent elderly people living in the community or in institutions. Age Ageing. 2007 May;36(3):298-303. doi: 10.1093/ageing/afm026. Epub 2007 Mar 24. PMID 17384419
- [Background] O'Connell S, Palmer R, Withers K, Saha N, Puntoni S, Carolan-Rees G; PROMs, PREMs and Effectiveness Programme. Requirements for the collection of electronic PROMS either "in clinic" or "at home" as part of the PROMs, PREMs and Effectiveness Programme (PPEP) in Wales: a feasibility study using a generic PROM tool. Pilot Feasibility Stud. 2018 Jul 4;4:90. doi: 10.1186/s40814-018-0282-8. eCollection 2018. PMID 29997899
- [Background] Duncanson E, Bennett PN, Viecelli A, Dansie K, Handke W, Tong A, Palmer S, Jesudason S, McDonald SP, Morton RL; Symptom monitoring WIth Feedback Trial (SWIFT) Investigators. Feasibility and acceptability of e-PROMs data capture and feedback among patients receiving haemodialysis in the Symptom monitoring WIth Feedback Trial (SWIFT) pilot: protocol for a qualitative study in Australia. BMJ Open. 2020 Nov 6;10(11):e039014. doi: 10.1136/bmjopen-2020-039014. PMID 33158824
- [Background] Anderson KO, Palos GR, Mendoza TR, Cleeland CS, Liao KP, Fisch MJ, Garcia-Gonzalez A, Rieber AG, Nazario LA, Valero V, Hahn KM, Person CL, Payne R. Automated pain intervention for underserved minority women with breast cancer. Cancer. 2015 Jun 1;121(11):1882-90. doi: 10.1002/cncr.29204. Epub 2015 Feb 24. PMID 25711974
- [Background] Adam R, Burton CD, Bond CM, de Bruin M, Murchie P. Can patient-reported measurements of pain be used to improve cancer pain management? A systematic review and meta-analysis. BMJ Support Palliat Care. 2017 Dec;7(4):0. doi: 10.1136/bmjspcare-2016-001137. Epub 2016 Nov 22. PMID 27879472
- [Background] Mooney KH, Beck SL, Friedman RH, Farzanfar R, Wong B. Automated monitoring of symptoms during ambulatory chemotherapy and oncology providers' use of the information: a randomized controlled clinical trial. Support Care Cancer. 2014 Sep;22(9):2343-50. doi: 10.1007/s00520-014-2216-1. Epub 2014 Apr 1. PMID 24687538
- [Background] Vasey B, Ursprung S, Beddoe B, Taylor EH, Marlow N, Bilbro N, Watkinson P, McCulloch P. Association of Clinician Diagnostic Performance With Machine Learning-Based Decision Support Systems: A Systematic Review. JAMA Netw Open. 2021 Mar 1;4(3):e211276. doi: 10.1001/jamanetworkopen.2021.1276. PMID 33704476
- [Background] Adler-Milstein J, Chen JH, Dhaliwal G. Next-Generation Artificial Intelligence for Diagnosis: From Predicting Diagnostic Labels to "Wayfinding". JAMA. 2021 Dec 28;326(24):2467-2468. doi: 10.1001/jama.2021.22396. No abstract available. PMID 34882190
- [Background] Barrachina-Fernandez M, Maitin AM, Sanchez-Avila C, Romero JP. Wearable Technology to Detect Motor Fluctuations in Parkinson's Disease Patients: Current State and Challenges. Sensors (Basel). 2021 Jun 18;21(12):4188. doi: 10.3390/s21124188. PMID 34207198
- [Background] Khalil H, Bell B, Chambers H, Sheikh A, Avery AJ. Professional, structural and organisational interventions in primary care for reducing medication errors. Cochrane Database Syst Rev. 2017 Oct 4;10(10):CD003942. doi: 10.1002/14651858.CD003942.pub3. PMID 28977687
- [Background] Beaudouin, Valérie and Bloch, Isabelle and Bounie, David and Bounie, David and Clémençon, Stéphan and d'Alché-Buc, Florence and Eagan, James and Maxwell, Winston and Mozharovskyi, Pavlo and Parekh, Jayneel, Flexible and Context-Specific AI Explainability: A Multidisciplinary Approach (March 23, 2020). Available at SSRN: https://ssrn.com/abstract=3559477 or http://dx.doi.org/10.2139/ssrn.3559477
- [Derived] Havreng-Thery C, Fouchard A, Denis F, Veyron JH, Belmin J. Cost-Effectiveness Analysis of a Machine Learning-Based eHealth System to Predict and Reduce Emergency Department Visits and Unscheduled Hospitalizations of Older People Living at Home: Retrospective Study. JMIR Form Res. 2025 Apr 11;9:e63700. doi: 10.2196/63700. PMID 40215100
- [Derived] Veyron JH, Deparis F, Al Zayat MN, Belmin J, Havreng-Thery C. Postimplementation Evaluation in Assisted Living Facilities of an eHealth Medical Device Developed to Predict and Avoid Unplanned Hospitalizations: Pragmatic Trial. J Med Internet Res. 2024 Dec 10;26:e55460. doi: 10.2196/55460. PMID 39657177
- [Derived] Belmin J, Villani P, Gay M, Fabries S, Havreng-Thery C, Malvoisin S, Denis F, Veyron JH. Real-world Implementation of an eHealth System Based on Artificial Intelligence Designed to Predict and Reduce Emergency Department Visits by Older Adults: Pragmatic Trial. J Med Internet Res. 2022 Sep 8;24(9):e40387. doi: 10.2196/40387. PMID 35921685